CLINICAL TRIAL: NCT04153825
Title: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) and Interferential Currents (IFC) on Central Sensitization in Patients With Knee Osteoarthritis: Randomized Clinical Trial
Brief Title: Comparison of Effectiveness of Two Different Electrotherapy Agents on Central Sensitization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turkish League Against Rheumatism (Other)
Responsible Party: Principal Investigator, Şahide Eda Almaz, Principal Investigator, MD, Turkish League Against Rheumatism
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRASD1
Record Dates: First submitted 2019-10-30; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Physical therapy modalities; Osteoarthritis knee; Central nervous system sensitization; Pain; Electric Stimulation Therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Transcutaneous Electric Nerve Stimulation; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Active TENS Group (Active Comparator): Ten sessions of active conventional TENS and hydrocollator hot-pack.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Other: Hydrocollator hot-pack
- Active IFC Group (Active Comparator): Ten sessions of active interferential current and hydrocollator hot-pack.
  Interventions: Device: Interferential Current; Other: Hydrocollator hot-pack
- Sham TENS Group (Sham Comparator): Ten sessions of sham TENS and hydrocollator hot-pack.
  Interventions: Other: Hydrocollator hot-pack; Device: Sham transcutaneous Electrical Nerve Stimulation
- Sham IFC Group (Sham Comparator): Ten sessions of sham IFC and hydrocollator hot-pack.
  Interventions: Other: Hydrocollator hot-pack; Device: Sham interferential Current

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Electrodes are placed around painful regions determined by the patient as patients are in the sitting position with the knees extended. The device is set at pulse duration of 50 to 80 μs; pulse frequency of 50 to 100 Hz; low-intensity (paraesthesia, not painful). The patient wears TENS for a 20-minute duration for each knee.
  Other Names: TENS
  Arms: Active TENS Group
Device: Interferential Current — Electrodes are placed diagonally around the painful areas defined by the patient, with the patient in the sitting position with the knees extended. The device is set at carrier frequency 4000 Hz, amplitude modulated frequency (AMF) 100 Hz, scanning frequency 50 Hz, scanning mode 1: 1 s. The patient wears ICF for a 20-minute duration for each knee.
  Other Names: IFC
  Arms: Active IFC Group
Other: Hydrocollator hot-pack — The hot-pack (at a surface temperature of almost 42 °C) is administered on knees while patients are in sitting position with the knees extended. Every session includes 20 minutes of hot-pack for each knee.
Device: Sham transcutaneous Electrical Nerve Stimulation — Electrodes are placed around painful regions determined by the patient as patients are in the sitting position with the knees extended.TENS unit in place but not turned on.The patient wears TENS for a 20-minute duration for each knee.
  Other Names: Sham TENS
  Arms: Sham TENS Group
Device: Sham interferential Current — Electrodes are placed diagonally around the painful areas defined by the patient, with the patient in the sitting position with the knees extended. IFC unit in place but not turned on.The patient wears ICF for a 20-minute duration for each knee.
  Other Names: Sham IFC
  Arms: Sham IFC Group

SUMMARY:
The aim of this study is to compare the efficacy of transcutaneous electrical nerve stimulation (TENS), interferential currents (IFCs) and sham devices in improving central sensitization (CS) findings, including pressure pain thresholds, pain catastrophizing, depression, and kinesiophobia in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Knee OA, which is the most frequently encountered type of OA is a leading cause of disability and chronic pain. CS is as important as nociceptive component in the pathogenesis of OA-related pain. Therefore, the necessary interventions for CS should be also considered when deciding the treatment protocol.TENS and IFC have been safely and commonly employed in the conservative treatment of knee OA. However, there are limited and inconsistent data concerning the impact of these modalities on CS component of pain.Therefore, the aim of this study is to investigate whether these agents are effective on CS and they are superior to each other.

ELIGIBILITY:
Inclusion Criteria:

40 to 75 years of age, Having bilateral knee OA radiologically with a Kellgren-Lawrence grade of 2 or 3.

Reporting knee pain of more than 3 on the visual analog scale (VAS) over the last 6 months Being unfamiliar with TENS and IFC use

-

Exclusion Criteria:

1. Having the history of any contraindication for electrotherapy (pacemakers, epilepsy, dermatological conditions, abnormal sensation in the knees, pregnancy),
2. Having a knee surgery or intra-articular corticosteroid or hyaluronic acid injection within 6 months.
3. Taking any drugs acting on the nervous system such as anticonvulsants, antidepressants, myorelaxants, or opioid drugs in the study period.
4. Having fibromyalgia, inflammatory rheumatologic, severe psychological disorders -

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Pressure-pain thresholds | Change from baseline pressure-pain thresholds at 2 weeks and at 12 weeks
  Pressure pain thresholds is measured on the knee (M. Vastus Medialis) and on the upper part of the homolateral arm (lateral part of M. Deltoideus, 10 cm below acromion) using a pressure algometer. The pressure is raised at a rate of almost 1 kg/s, until the patient first notifies that the pressure sensation changes to a pain sensation.
Tampa Scale of Kinesiophobia | Change from baseline kinesiophobia scores at 2 weeks and at 12 weeks
  Tampa Scale contains 17 parts that measure anxiety and fear related to movement. The total score ranges between 17-68 points. Higher scores represent higher grades of kinesiophobia.
Beck Depression Inventory (BDI) | Change from baseline BDI scores at 2 weeks and at 12 weeks.
  Beck Depression Inventory is a 21-item questionnaire that examines the characteristic symptoms of depression.
Pain catastrophizing scale (PCS) | Change from baseline PCS scores at 2 weeks and at 12 weeks.
  PCS consists of 13 items in three subscales (rumination, helplessness, and magnification). Higher final score indicates more catastrophic thinking related to pain.

SECONDARY OUTCOMES:
Age | Baseline
  years
Gender | Baseline
  female/male
Height | Baseline
  centimeter (cm)
Weight | Baseline
  kilogram (kg)
Comorbidity | Baseline
  self reported
Visual analogue scale (VAS) | Change from baseline, at 2 weeks and at 12 weeks
  VAS ranging levels from 0 (no pain) to 10 (maximal pain).
Western Ontario and McMaster University (WOMAC) Index. | Change from baseline, at 2 weeks and at 12 weeks
  There are three subscales with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Timed Up and Go Test (TUG) | Change from baseline, at 2 weeks and at 12 weeks
  Timed up and go test is used to assess mobility which recorded the time of rising from a back-rest chair, walking at a normal pace 3 meters, turning, walking back to the chair, and sitting recumbently. In one minute durations, each participant will perform the test three times and this time will be recorded in seconds.
Five Times Sit to Stand Test | Change from baseline, at 2 weeks and at 12 weeks
  The participant is asked to sit-to-stand action from a standard chair five times as quickly as possible, and the time taken to complete is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Şahide E Almaz, MD, Principal Investigator — Turkish League Against Rheumatism; Hatice Bodur, Professor, Study Director — Turkish League Against Rheumatism; Aslı Çalışkan Uçkun, MD, Study Chair — Turkish League Against Rheumatism; Filiz Acar Sivas, Professor, Study Chair — Turkish League Against Rheumatism; Fatma G Yurdakul, MD, Study Chair — Turkish League Against Rheumatism
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All the collected data will be shared with investigators of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code